CLINICAL TRIAL: NCT02195999
Title: Assessment of Cardiopulmonary Function in Duchenne Muscular Dystrophy
Acronym: CPI
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: CureDuchenne (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300420
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Magnetic Resonance Spectroscopy; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with DMD: Magnetic Resonance Imaging is a non-invasive method to determine ventricular size, volumes, mass, and ejection fraction.
  Pulmonary Function testing (PFT) are a series of non-invasive breathing tests that characterize respiratory muscle function, as well as lung compliance and physiology.
  Metabolic exercise testing using stationary bicycle (exercise capacity and MVO2) evaluates global cardiopulmonary functional status.
  Echocardiogram with multiple-echo Dixon method helps to assess cross-sectional and longitudinal variations in myocardial structure.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Other: Pulmonary Function Testing (PFT); Other: Metabolic Exercise Testing using stationary bicycle; Other: Echocardiogram

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — It is a non-invasive method to determine ventricular size, volumes, mass, and ejection fraction.
Other: Pulmonary Function Testing (PFT) — It is non-invasive breathing tests that characterize respiratory muscle function, as well as lung compliance and physiology.
Other: Metabolic Exercise Testing using stationary bicycle — Metabolic exercise testing, including assessment of exercise capacity and MVO2, evaluates global cardiopulmonary functional status. This is performed with the use of a stationary bicycle.
Other: Echocardiogram — The echocardiogram performed with the multiple-echo Dixon method helps to assess participants cross-sectionally and longitudinally for variations and changes in myocardial structure.
  Other Names: Multiple-echo Dixon

SUMMARY:
This study seeks to develop and validate non-invasive assessments of cardiac and respiratory muscles with magnetic resonance imaging (MRI) to better predict the natural disease progression of Duchenne muscular dystrophy (DMD) in affected individuals over time, as well as determine whether peripheral skeletal muscle dysfunction can predict cardiopulmonary dysfunction. The central hypothesis is that non-invasive MRI measures of the heart, muscle, and peripheral skeletal muscles can sensitively predict future cardiopulmonary decline.

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) of the heart and breathing muscles, special breathing tests (called pulmonary function testing), special exercise tests (using a stationary bike), and possibly an echocardiogram (ultrasound of the heart, commonly known as an "echo") will be completed up to 4 times per year for up to 4 years. Most participants will complete testing once or twice each year; however, some participants will be asked to repeat some of the tests twice during each visit.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 5-15 years old at the time of enrollment
* Diagnosed with DMD (as defined by parent project)
* Written parental informed consent (and assent where appropriate) before any study procedures take place

Exclusion Criteria:

* Contraindication to an MRI examination
* Presence of a secondary condition that impacts muscle function or metabolism, that leads to developmental delay or impaired motor control, or that is not stable
* Participant is unable to comply with study requirements
* Congenital structural abnormality of the heart, repaired or unrepaired
* Clinically contraindicated participation

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: As the focus of this study is on validating novel measures of cardiac and respiratory function in individuals with DMD, this study will utilize a single-group design with up to 60 males with DMD between 5 and 15 years old upon entry to the study. The participant selection is limited to children since the detrimental effects of DMD begin in early childhood, and the life expectancy of these boys is shortened to the early- to mid-20s. Only males will be eligible to participate in the study because DMD is an X-linked recessive genetic disorder that only leads to the characteristic disease in males. Although females may be carriers, they do not exhibit the same phenotype as males.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance (MRI) T2 and Magnetic Resonance Spectroscopy (MRS) | up to 4 years
  The MRI T2 and MRS will be used as a noninvasive marker of myocardial damage/inflammation of participants of this study as an early detection for DMD.

SECONDARY OUTCOMES:
Pulmonary Function Testing (PFT) | up to 4 years
  Non-invasive breathing tests that characterize respiratory muscle function, as well as lung compliance and physiology.
Metabolic Exercise Testing (exercise capacity and MVO2) | up to 4 years
  With the use of metabolic exercise testing, the aim is to correlate changes in cardiopulmonary function with decline in peripheral skeletal muscle function in individuals with DMD. Metabolic exercise testing includes measuring exercise capacity and maximum oxygen consumption (MVO2).
Multiple-echo Dixon | up to 4 years
  The echocardiogram performed with the multiple-echo Dixon method helps to assess participants cross-sectionally and longitudinally for variations and changes in myocardial structure. This method and MRS will also be used for fat fraction determination.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Byrne, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- Clinical and Translational Research Building, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No